CLINICAL TRIAL: NCT00552175
Title: A Superiority Study of LY248686 Versus Placebo in the Treatment of Patients With Diabetic Peripheral Neuropathic Pain
Brief Title: A Study for the Treatment of Diabetic Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Shionogi (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12191; 0715N0831 (Other: Shionogi & Co., Ltd); F1J-JE-HMFX (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Results first posted 2010-04-13 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-03

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Duloxetine 60 (Experimental): duloxetine 60 milligram (mg) taken orally every day
  Interventions: Drug: Duloxetine hydrochloride - 60 mg
- Duloxetine 40 (Experimental): Duloxetine 40 mg taken orally every day
  Interventions: Drug: Duloxetine hydrochloride - 40 mg
- Placebo (Placebo Comparator): placebo comparator taken orally every day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Duloxetine hydrochloride - 40 mg — duloxetine 40 mg taken orally every day
  Other Names: LY248686; Cymbalta
  Arms: Duloxetine 40
Drug: placebo — placebo taken orally every day
  Arms: Placebo
Drug: Duloxetine hydrochloride - 60 mg — duloxetine 60 mg taken orally every day
  Other Names: LY248686; Cymbalta
  Arms: Duloxetine 60

SUMMARY:
The purpose of the study is to determine if duloxetine can help patients with painful diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pain due to bilateral peripheral neuropathy induced by type 1 or 2 diabetes mellitus. The pain must have been present for at least 6 months and be evaluable in feet, legs, or hands.
* Participants with hemoglobin A1c (HbA1c) less than or equal to 9.0 percent at Visit 1.
* Participants in whom HbA1c had been measured 42-70 days before Visit 1 and subsequent HbA1c levels have been within +/- 1.0 percent of the level at Visit 1.
* Participants with a mean of the 24-hour average pain severity scores (round off to a whole number) of 4 or higher, as calculated from the patient diary for 7 days immediately before Visit 2

Exclusion Criteria:

* Participants who have undergone renal transplant or who are currently on renal dialysis.
* Participants who have a history requiring pharmacotherapy within the past year or current history of psychiatric disease, such as mania, bipolar disorder, depression, anxiety disorder, or eating disorder.
* Participants with hypertension with poor control of blood pressure (systolic blood pressure greater than or equal to 180 millimeters of mercury (mmHg) or diastolic blood pressure greater than or equal to 110 mmHg
* Participants with alanine transaminase (ALT) or aspartate transaminase (AST) greater than or equal to 100 Units per Liter (U/L) at Visit 1.
* Participants unable to discontinue prohibited concomitant drugs or concomitant therapies after Visit 1.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2007-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) OR 1-317-615-4559 Mon-Fri 9 AM-5 PM Eastern time (UTC/GMT-5 hours,EST), Study Director — Eli Lilly and Company
Locations (25):
- Japan (25):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aomori
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukui
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gunma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT -5 hours, ETS), or speak with your personal physician, Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagoshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyagi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niigata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT -5 hours, ETS), or speak with your personal physician, Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ōita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tochigi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toyama

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Full Analysis Set Population consisted of all randomized patients who had at least one post-baseline measure of the primary efficacy variable.
Groups:
- Duloxetine 40 mg: Duloxetine 40 milligrams (mg) taken orally every day
- Duloxetine 60 mg: Duloxetine 60 milligrams (mg) taken orally every day
Period: Overall Study
Arm/Group | Placebo | Duloxetine 40 mg | Duloxetine 60 mg
Started | 167 | 86 | 86
Full Analysis Set Population | 167 | 85 | 86
Completed | 150 | 73 | 72
Not Completed | 17 | 13 | 14
Not completed — Lack of Efficacy | 2 | 0 | 1
Not completed — Adverse Event | 9 | 9 | 10
Not completed — Withdrawal by Subject | 2 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Entry Criteria Not Met | 1 | 1 | 0
Not completed — Reason Not Specified | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Duloxetine 40 mg | Duloxetine 60 mg | Total
Number analyzed (Participants) | 167 | 85 | 86 | 338
Age Continuous [Mean (Standard Deviation); unit: years] | 60.8 (9.2) | 62.1 (9.3) | 59.7 (12.1) | 60.8 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 20 | 24 | 82
  Male | 129 | 65 | 62 | 256
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 167 | 85 | 86 | 338
Region of Enrollment [Number; unit: participants]
  Japan | 167 | 85 | 86 | 338
Duration of Diabetes [Number; unit: participants]
  <5 years | 33 | 20 | 16 | 69
  5 - 10 years | 32 | 18 | 14 | 64
  >= 10 years | 97 | 47 | 56 | 200
  Unknown | 5 | 0 | 0 | 5
Type of Diabetes [Number; unit: participants]
  Type I | 8 | 5 | 4 | 17
  Type II | 159 | 80 | 82 | 321
Beck Depression Inventory-II (BDI-II) [Mean (Standard Deviation); unit: units on a scale] — A 21-item, patient-completed questionnaire to assess characteristics of depression. Each of the 21 items corresponding to a symptom of depression is summed to give a single score. There is a four-point scale for each item ranging from 0 to 3. Total score ranges from 0 (no depression) to 63 (severe depression).
  units on a scale | 8.8 (6.8) | 9.4 (8.8) | 9.4 (7.2) | 9.1 (7.4)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/square meters (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms/square meters (kg/m^2) | 23.90 (3.70) | 23.27 (3.67) | 24.20 (3.50) | 23.82 (3.65)
Brief Pain Inventory (BPI) Interference Scores [Mean (Standard Deviation); unit: units on a scale] — The Interference scores range from 0 (does not interfere) to 10 (completely interferes). There are 7 questions assessing the interference of pain in the past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Each question has total scores ranging from 0 to 10.
  units on a scale
    General Activity | 4.4 (2.4) | 4.5 (2.7) | 4.5 (2.4) | 4.5 (2.5)
    Mood | 4.2 (2.4) | 3.9 (2.5) | 4.2 (2.5) | 4.1 (2.5)
    Walking Ability | 4.0 (2.6) | 4.4 (2.8) | 4.3 (2.5) | 4.2 (2.6)
    Normal Work | 3.7 (2.7) | 3.9 (2.6) | 4.3 (2.5) | 3.9 (2.6)
    Relation to People | 2.6 (2.5) | 2.7 (2.7) | 2.9 (2.4) | 2.7 (2.5)
    Sleep | 3.9 (2.7) | 4.0 (2.8) | 4.3 (2.7) | 4.0 (2.7)
    Enjoyment of Life | 3.5 (2.5) | 3.7 (2.7) | 4.0 (2.5) | 3.7 (2.6)
    Average of Interference Scores | 3.75 (2.15) | 3.88 (2.25) | 4.09 (2.13) | 3.87 (2.17)
Brief Pain Inventory (BPI) Severity Scores [Mean (Standard Deviation); unit: units on a scale] — A self-reported scale that measures the severity of pain and the interference of pain on function. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). There are 4 questions assessing worst pain, least pain, and average pain in the past 24 hours, and the pain right now. Each question has a total range of scores from 0 to 10.
  units on a scale
    Worst Pain | 6.7 (1.4) | 6.5 (1.4) | 6.6 (1.5) | 6.6 (1.4)
    Least Pain | 4.1 (1.8) | 4.0 (1.8) | 4.2 (1.6) | 4.1 (1.8)
    Average Pain | 5.6 (1.3) | 5.6 (1.3) | 5.7 (1.3) | 5.6 (1.3)
    Pain Right Now | 5.1 (1.7) | 5.2 (1.8) | 5.3 (1.4) | 5.2 (1.7)
Duration of Diabetic Neuropathy [Mean (Standard Deviation); unit: years] | 4.21 (4.44) | 4.58 (3.90) | 4.16 (3.67) | 4.29 (4.11)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 164.13 (8.65) | 163.63 (8.78) | 164.02 (7.32) | 163.98 (8.34)
Weekly Means of 24-Hour Average Pain, Worst Pain, and Night Pain Diary Scores [Mean (Standard Deviation); unit: units on a scale] — 24-hour average pain severity scores recorded in a diary daily on an 11-point numerical rating scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). The 11-point numerical rating scale was also used for assessment of night pain and worst pain each day, and evaluated as weekly means. Total scores for each pain assessment (average, worst, night) range from 0 to 10.
  units on a scale
    Average Pain Score | 5.78 (1.17) | 5.79 (1.23) | 5.76 (1.17) | 5.78 (1.18)
    Worst Pain Score | 6.66 (1.25) | 6.54 (1.33) | 6.61 (1.33) | 6.62 (1.29)
    Night Pain Score | 5.5 (1.49) | 5.55 (1.64) | 5.69 (1.54) | 5.56 (1.54)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 64.52 (11.93) | 62.72 (13.35) | 65.08 (10.23) | 64.21 (11.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 12 in Average Pain Severity Rating Using Diaries for the Combined Duloxetine Arms (40 mg + 60 mg)
Description: Average pain severity was measured using an 11-point numerical rating scale, collected by diaries and expressed as weekly mean. The scale is a self-reported instrument that measures the severity of pain based on the average pain over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline, 12 weeks
Population: Patients in the Full Analysis Set Population who had a post-baseline measurement in the variable being presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Duloxetine 40 mg and 60 mg Combined: Duloxetine 40 milligrams (mg) taken orally every day, and Duloxetine 60 mg taken orally every day.
Arm/Group | Placebo | Duloxetine 40 mg and 60 mg Combined
Number analyzed (Participants) | 167 | 171
units on a scale | -1.61 (0.18) | -2.47 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 40 mg and 60 mg Combined; The primary objective and primary efficacy analysis for the study was the analysis between the combined duloxetine arms and placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Covariates: Baseline value of average pain score, type of Diabetes, Duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.87, 95% CI 2-sided [-1.17 to -0.56], Standard Error of Mean 0.15 — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo

2. Secondary Outcome: Change From Baseline at Week 12 in Average Pain Severity Rating Score Using Diaries
Description: as for outcome 1
Time Frame: Baseline, 12 weeks
Population: Patients in the Full Analysis Set Population who had a post-baseline measurement in the variable being presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine 40 mg | Duloxetine 60 mg
Number analyzed (Participants) | 167 | 85 | 86
units on a scale | -1.61 (0.19) | -2.41 (0.21) | -2.53 (0.21)

3. Secondary Outcome: Change From Baseline at Week 12 in Worst Pain Severity Score and Night Pain Severity Score Using Diaries for the Combined Duloxetine Arms (40 mg + 60 mg)
Description: Pain severity for worst pain and night pain as measured by an 11-point numerical rating scale, collected by diaries and expressed as weekly means. A self-reported scale that measures the severity of pain based on the worst pain and night pain experienced over the past 24-hours. The worst pain and night pain severity scores each range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline, 12 weeks
Population: Patients in the Full Analysis Set Population who had a post-baseline measurement in the variable being presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine 40 mg and 60 mg Combined
Number analyzed (Participants) | 167 | 171
units on a scale
  Worst Pain | -1.55 (0.19) | -2.51 (0.19)
  Night Pain | -1.56 (0.19) | -2.39 (0.19)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 40 mg and 60 mg Combined; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for Worst Pain; Covariates: Baseline value of worst pain score, type of Diabetes, Duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.96, 95% CI 2-sided [-1.27 to -0.64] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Duloxetine 40 mg and 60 mg Combined; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for Night Pain; Covariates: Baseline value of night pain score, type of Diabetes, Duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.83, 95% CI 2-sided [-1.15 to -0.51] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo

4. Secondary Outcome: Change From Baseline at Week 12 in Worst Pain Severity Score and Night Pain Severity Score Using Diaries
Description: as for outcome 3
Time Frame: Baseline, Week 12
Population: Patients in the Full Analysis Set Population who had a post-baseline measurement in the variable being presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine 40 mg | Duloxetine 60 mg
Number analyzed (Participants) | 167 | 85 | 86
units on a scale
  Worst Pain | -1.55 (0.19) | -2.42 (0.22) | -2.59 (0.22)
  Night Pain | -1.56 (0.19) | -2.33 (0.22) | -2.45 (0.23)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 40 mg; Worst Pain analysis; Test type: Superiority or Other; Mixed Models Analysis; Covariates: Baseline value of worst pain score, type of diabetes, and duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.87, 95% CI 2-sided [-1.26 to -0.49] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Duloxetine 60 mg; Worst Pain analysis; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 4, analysis 1]; Least Squares Mean Difference = -1.05, 95% CI 2-sided [-1.43 to -0.66] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 40 mg; Night Pain analysis; Test type: Superiority or Other; Mixed Models Analysis; Covariates: Baseline value of night pain score, type of diabetes, and duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.78, 95% CI 2-sided [-1.17 to -0.39] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 60 mg; Night Pain analysis; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 4, analysis 3]; Least Squares Mean Difference = -0.89, 95% CI 2-sided [-1.28 to -0.5] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo

5. Secondary Outcome: Patient Global Impression of Improvement Scale at Week 12 in Combined Duloxetine Arms (40 mg + 60 mg)
Description: A scale that measures the patient's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from 1 (very much better) to 7 (very much worse).
Time Frame: Week 12
Population: Patients in the Full Analysis Set Population who had a post-baseline measurement in the variable being presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine 40 mg and 60 mg Combined
Number analyzed (Participants) | 165 | 169
units on a scale | 3.18 (0.12) | 2.53 (0.12)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 40 mg and 60 mg Combined; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.65, 95% CI 2-sided [-0.85 to -0.44] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo

6. Secondary Outcome: Patient Global Impression of Improvement Scale at Week 12
Description: as for outcome 5
Time Frame: Week 12
Population: Patients in the Full Analysis Set Population who had a post-baseline measurement in the variable being presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine 40 mg | Duloxetine 60 mg
Number analyzed (Participants) | 165 | 84 | 85
units on a scale | 3.18 (0.12) | 2.53 (0.14) | 2.52 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 40 mg; Test type: Superiority or Other; Mixed Models Analysis; Covariates: Baseline value of average pain score, type of diabetes, and duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.65, 95% CI 2-sided [-0.9 to -0.39] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.65, 95% CI 2-sided [-0.91 to -0.4] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo

7. Secondary Outcome: Change From Baseline in Brief Pain Inventory Severity Scores at Week 12 for the Combined Duloxetine Arms (40 mg + 60 mg)
Description: A self-reported scale that measures the severity of pain. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). There are 4 questions assessing worst pain, least pain, and average pain in the past 24 hours, and the pain right now. Each question has a total range of scores from 0 to 10.
Time Frame: Baseline, Week 12
Population: Patients in the Full Analysis Set Population who had a post-baseline measurement in the variable being presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine 40 mg and 60 mg Combined
Number analyzed (Participants) | 165 | 169
units on a scale
  Worst Pain | -1.62 (0.21) | -2.59 (0.21)
  Least Pain | -1.13 (0.21) | -1.98 (0.21)
  Average Pain | -1.54 (0.2) | -2.54 (0.2)
  Pain Right Now | -1.67 (0.22) | -2.59 (0.22)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 40 mg and 60 mg Combined; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for Worst Pain; [statistical method as in outcome 3, analysis 1]; Least Squares Mean Difference = -0.98, 95% CI 2-sided [-1.34 to -0.61] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Duloxetine 40 mg and 60 mg Combined; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for Least Pain; Covariates: Baseline value of least pain score, type of Diabetes, Duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.85, 95% CI 2-sided [-1.21 to -0.48] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 40 mg and 60 mg Combined; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for Average Pain; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -1, 95% CI 2-sided [-1.33 to -0.67] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 40 mg and 60 mg Combined; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for Pain Right Now; Covariates: Baseline value of pain right now score, type of Diabetes, Duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.92, 95% CI 2-sided [-1.29 to -0.54] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo

8. Secondary Outcome: Change From Baseline in Brief Pain Inventory Severity Scores at Week 12
Description: as for outcome 7
Time Frame: Baseline, Week 12
Population: Patients in the Full Analysis Set Population who had a post-baseline measurement in the variable being presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine 40 mg | Duloxetine 60 mg
Number analyzed (Participants) | 165 | 84 | 85
units on a scale
  Worst Pain | -1.62 (0.21) | -2.51 (0.25) | -2.68 (0.25)
  Least Pain | -1.13 (0.21) | -1.92 (0.25) | -2.04 (0.25)
  Average Pain | -1.55 (0.2) | -2.53 (0.23) | -2.56 (0.23)
  Pain Right Now | -1.67 (0.22) | -2.55 (0.25) | -2.62 (0.26)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 40 mg; Worst Pain Score analysis; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 4, analysis 1]; Least Squares Mean Difference = -0.89, 95% CI 2-sided [-1.34 to -0.44] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Duloxetine 60 mg; Worst Pain Score analysis; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 4, analysis 1]; Least Squares Mean Difference = -1.06, 95% CI 2-sided [-1.51 to -0.62] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 40 mg; Least Pain Score analysis; Test type: Superiority or Other; Mixed Models Analysis; Covariates: Baseline value of least pain score, type of diabetes, and duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.78, 95% CI 2-sided [-1.23 to -0.33] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 60 mg; Least Pain Score analysis; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 8, analysis 3]; Least Mean Squares Difference = -0.91, 95% CI 2-sided [-1.36 to -0.46] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Duloxetine 40 mg; Average Pain Score analysis; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.98, 95% CI 2-sided [-1.39 to -0.58] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 6: Comparison: Placebo vs Duloxetine 60 mg; Average Pain Score analysis; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 6, analysis 1]; Least Squares Mean Difference = -1.01, 95% CI 2-sided [-1.41 to -0.61] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 7: Comparison: Placebo vs Duloxetine 40 mg; Pain Right Now Score analysis; Test type: Superiority or Other; Mixed Models Analysis; Covariates: Baseline value of pain right now score, type of diabetes, and duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.88, 95% CI 2-sided [-1.35 to -0.41] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 8: Comparison: Placebo vs Duloxetine 60 mg; Pain Right Now Score analysis; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 8, analysis 7]; Least Squares Mean Difference = -0.95, 95% CI 2-sided [-1.41 to -0.48] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo

9. Secondary Outcome: Change From Baseline in Brief Pain Inventory Interference Scores at Week 12 for the Combined Duloxetine Arms (40 mg + 60 mg)
Description: The Interference scores range from 0 (does not interfere) to 10 (completely interferes). There are 7 questions assessing the interference of pain in the past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Each question has a total range of scores from 0 to 10.
Time Frame: Baseline, Week 12
Population: Patients in the Full Analysis Set Population who had a post-baseline measurement in the variable being presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine 40 mg and 60 mg Combined
Number analyzed (Participants) | 165 | 169
units on a scale
  General Activity | -1.88 (0.24) | -2.29 (0.24)
  Mood | -1.91 (0.24) | -2.28 (0.24)
  Walking Ability | -1.82 (0.23) | -2.31 (0.23)
  Normal Work | -1.49 (0.23) | -1.86 (0.23)
  Relation to People | -0.77 (0.23) | -1.32 (0.23)
  Sleep | -1.69 (0.24) | -2.15 (0.24)
  Enjoyment of Life | -1.59 (0.23) | -2.15 (0.23)
  Average of Interference Scores | -1.56 (0.2) | -2.04 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 40 mg and 60 mg Combined; Test type: Superiority or Other; p = 0.0676, Mixed Models Analysis — P-value for General Activity; Covariates: Baseline value of general activity score, type of Diabetes, Duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.41, 95% CI 2-sided [-0.85 to 0.03] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Duloxetine 40 mg and 60 mg Combined; Test type: Superiority or Other; p = 0.0933, Mixed Models Analysis — P-value for Mood; Covariates: Baseline value of mood score, type of Diabetes, Duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.37, 95% CI 2-sided [-0.8 to 0.06] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 40 mg and 60 mg Combined; Test type: Superiority or Other; p = 0.0228, Mixed Models Analysis — P-value for Walking Ability; Covariates: Baseline value of walking ability score, type of Diabetes, Duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.49, 95% CI 2-sided [-0.91 to -0.07] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 40 mg and 60 mg Combined; Test type: Superiority or Other; p = 0.0783, Mixed Models Analysis — P-value for Normal Work; Covariates: Baseline value of normal work score, type of Diabetes, Duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.38, 95% CI 2-sided [-0.8 to 0.04] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Duloxetine 40 mg and 60 mg Combined; Test type: Superiority or Other; p = 0.0076, Mixed Models Analysis — P-value for Relation to People; Covariates: Baseline value of relation to people score, type of Diabetes, Duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.55, 95% CI 2-sided [-0.96 to -0.15] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 6: Comparison: Placebo vs Duloxetine 40 mg and 60 mg Combined; Test type: Superiority or Other; p = 0.0378, Mixed Models Analysis — P-value for Sleep; Covariates: Baseline value of sleep score, type of Diabetes, Duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.46, 95% CI 2-sided [-0.9 to -0.03] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 7: Comparison: Placebo vs Duloxetine 40 mg and 60 mg Combined; Test type: Superiority or Other; p = 0.0089, Mixed Models Analysis — P-value for Enjoyment of Life; Covariates: Baseline value of enjoyment of life score, type of Diabetes, Duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.56, 95% CI 2-sided [-0.98 to -0.14] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 8: Comparison: Placebo vs Duloxetine 40 mg and 60 mg Combined; Test type: Superiority or Other; p = 0.0095, Mixed Models Analysis — P-value for Average of Interference Scores; Covariates: Baseline value of average of interference scores, type of Diabetes, Duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.48, 95% CI 2-sided [-0.85 to -0.12] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo

10. Secondary Outcome: Change From Baseline in Brief Pain Inventory Interference Scores at Week 12
Description: as for outcome 9
Time Frame: Baseline, Week 12
Population: Patients in the Full Analysis Set Population who had a post-baseline measurement in the variable being presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine 40 mg | Duloxetine 60 mg
Number analyzed (Participants) | 165 | 84 | 85
units on a scale
  General Activity | -1.88 (0.24) | -2.48 (0.29) | -2.1 (0.29)
  Mood | -1.91 (0.24) | -2.18 (0.29) | -2.39 (0.29)
  Walking Ability | -1.82 (0.23) | -2.32 (0.28) | -2.31 (0.28)
  Normal Work | -1.49 (0.23) | -1.84 (0.28) | -1.9 (0.28)
  Relation to People | -0.77 (0.23) | -1.16 (0.27) | -1.49 (0.27)
  Sleep | -1.69 (0.24) | -2.26 (0.29) | -2.05 (0.29)
  Enjoyment of Life | -1.59 (0.23) | -1.96 (0.28) | -2.35 (0.28)
  Average of Interference Scores | -1.56 (0.2) | -2 (0.24) | -2.08 (0.24)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 40 mg; General Activity score analysis; Test type: Superiority or Other; Mixed Models Analysis; Covariates: Baseline value of general activity, type of diabetes, and duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.6, 95% CI 2-sided [-1.14 to -0.06] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Duloxetine 60 mg; General Activity score analysis; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 10, analysis 1]; Least Squares Mean Difference = -0.23, 95% CI 2-sided [-0.77 to 0.32] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 40 mg; Mood score analysis; Test type: Superiority or Other; Mixed Models Analysis; Covariates: Baseline value of mood score, type of diabetes, and duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.27, 95% CI 2-sided [-0.8 to 0.27] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 60 mg; Mood score analysis; Test type: Superiority or Other; Mixed Models Analysis; Covariates: Baseline value of mood score, type of diabetes, and duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.48, 95% CI 2-sided [-1.01 to 0.05] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Duloxetine 40 mg; Walking Ability score analysis; Test type: Superiority or Other; Mixed Models Analysis; Covariates: Baseline value of walking ability, type of diabetes, and duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.5, 95% CI 2-sided [-1.02 to 0.02] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 6: Comparison: Placebo vs Duloxetine 60 mg; Walking Ability score analysis; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 10, analysis 5]; Least Squares Mean Difference = -0.49, 95% CI 2-sided [-1.01 to 0.03] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 7: Comparison: Placebo vs Duloxetine 40 mg; Normal Work score analysis; Test type: Superiority or Other; Mixed Models Analysis; Covariates: Baseline value of normal work score, type of diabetes, and duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.35, 95% CI 2-sided [-0.86 to 0.16] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 8: Comparison: Placebo vs Duloxetine 60 mg; Normal Work score analysis; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 10, analysis 7]; Least Squares Mean Difference = -0.41, 95% CI 2-sided [-0.92 to 0.11] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 9: Comparison: Placebo vs Duloxetine 40 mg; Relation to People score analysis; Test type: Superiority or Other; Mixed Models Analysis; Covariates: Baseline value of relation to people, type of diabetes, and duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.39, 95% CI 2-sided [-0.89 to 0.11] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 10: Comparison: Placebo vs Duloxetine 60 mg; Relation to People score analysis; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 10, analysis 9]; Least Squares Mean Difference = -0.71, 95% CI 2-sided [-1.21 to -0.22] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 11: Comparison: Placebo vs Duloxetine 40 mg; Sleep score analysis; Test type: Superiority or Other; Mixed Models Analysis; Covariates: Baseline value of sleep score, type of diabetes, and duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.57, 95% CI 2-sided [-1.11 to -0.03] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 12: Comparison: Placebo vs Duloxetine 60 mg; Sleep score analysis; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 10, analysis 11]; Least Squares Mean Difference = -0.36, 95% CI 2-sided [-0.9 to 0.18] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 13: Comparison: Placebo vs Duloxetine 40 mg; Enjoyment of Life score analysis; Test type: Superiority or Other; Mixed Models Analysis; Covariates: Baseline value of enjoyment of life, type of diabetes, and duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.37, 95% CI 2-sided [-0.88 to 0.15] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 14: Comparison: Placebo vs Duloxetine 60 mg; Enjoyment of Life score analysis; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 10, analysis 13]; Least Squares Mean Difference = -0.76, 95% CI 2-sided [-1.27 to -0.24] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 15: Comparison: Placebo vs Duloxetine 40 mg; Average of Interference scores analysis; Test type: Superiority or Other; Mixed Models Analysis; Covariates: Baseline value of average of interference scores, type of diabetes, and duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.45, 95% CI 2-sided [-0.9 to 0] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 16: Comparison: Placebo vs Duloxetine 60 mg; Average of Interference scores analysis; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 10, analysis 15]; Least Squares Mean Difference = -0.52, 95% CI 2-sided [-0.97 to -0.07] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo

11. Secondary Outcome: Change From Baseline in Beck Depression Inventory-II (BDI-II) Total Score at Week 12 for the Combined Duloxetine Arms (40 mg + 60 mg)
Description: A 21-item, patient-completed questionnaire to assess characteristics of depression. Each of the 21 items corresponding to a symptom of depression is summed to give a single score. There is a four-point scale for each item ranging from 0 to 3. Total score ranges from 0 (no depression) to 63 (severe depression).
Time Frame: Baseline, Week 12
Population: Patients in the Full Analysis Set Population who had a post-baseline measurement in the variable being presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine 40 mg and 60 mg Combined
Number analyzed (Participants) | 165 | 169
units on a scale | -3.27 (0.64) | -3.37 (0.64)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 40 mg and 60 mg Combined; Test type: Superiority or Other; p = 0.8517, Mixed Models Analysis; Covariates: Baseline value of BDI-II, type of diabetes, and duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.11, 95% CI 2-sided [-1.22 to 1.01] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo

12. Secondary Outcome: Change From Baseline in Beck Depression Inventory-II (BDI-II) Total Score at Week 12
Description: as for outcome 11
Time Frame: Baseline, Week 12
Population: Patients in the Full Analysis Set Population who had a post-baseline measurement in the variable being presented.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Duloxetine 40 mg | Duloxetine 60 mg
Number analyzed (Participants) | 165 | 84 | 85
units on a scale | -3.28 (0.65) | -2.94 (0.76) | -3.83 (0.77)
Statistical Analysis 1: Comparison: Placebo vs Duloxetine 40 mg; Test type: Superiority or Other; Mixed Models Analysis; Covariates: Baseline value of BDI-II, type of diabetes, and duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = 0.34, 95% CI 2-sided [-1.03 to 1.71] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; Mixed Models Analysis; Covariates: Baseline value of BDI-II, type of diabetes, and duration of diabetic peripheral neuropathic pain (DPNP); Least Squares Mean Difference = -0.55, 95% CI 2-sided [-1.92 to 0.81] — Least Squares Mean Difference = Duloxetine 40 mg and 60 mg Combined minus Placebo

ADVERSE EVENTS:
Arm/Group | Placebo | Duloxetine 40 mg | Duloxetine 60 mg
Serious Adverse Events (participants affected / at risk) | 6/167 | 3/85 | 2/86
Other Adverse Events (participants affected / at risk) | 121/167 | 71/85 | 73/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=167) | Duloxetine 40 mg (N=85) | Duloxetine 60 mg (N=86)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tuberculous pleurisy (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urine albumin/creatinine ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Facial palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Thalamus haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Self injurious behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=167) | Duloxetine 40 mg (N=85) | Duloxetine 60 mg (N=86)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 4 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (9) | 6 (6) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 4 (5) | 7 (7)
Nausea (Gastrointestinal disorders) | 3 (3) | 10 (11) | 14 (17)
Stomach discomfort (Gastrointestinal disorders) | 4 (4) | 3 (4) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (5) | 5 (7)
Malaise (General disorders) | 3 (3) | 3 (3) | 6 (7)
Thirst (General disorders) | 3 (3) | 4 (4) | 4 (4)
Nasopharyngitis (Infections and infestations) | 24 (24) | 10 (11) | 14 (16)
Alanine aminotransferase increased (Investigations) | 6 (6) | 5 (5) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 5 (5) | 8 (8)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 4 (4) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 6 (6) | 6 (6) | 0 (0)
Blood glucose decreased (Investigations) | 7 (15) | 2 (4) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 4 (4) | 2 (2) | 5 (5)
Gamma-glutamyltransferase increased (Investigations) | 4 (4) | 2 (2) | 5 (5)
Glycosylated haemoglobin increased (Investigations) | 4 (4) | 1 (1) | 5 (5)
White blood cell count increased (Investigations) | 4 (4) | 4 (4) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (4)
Dizziness (Nervous system disorders) | 2 (3) | 6 (8) | 4 (4)
Headache (Nervous system disorders) | 6 (9) | 4 (4) | 2 (3)
Somnolence (Nervous system disorders) | 14 (14) | 16 (16) | 21 (23)
Eczema (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1) | 4 (4)

LIMITATIONS AND CAVEATS:
The protocol-specified primary analyses for this study were comparisons between combined duloxetine arms (40 mg + 60 mg) and placebo. The study was powered on combined duloxetine arms and statistical comparisons were not performed among single arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days